CLINICAL TRIAL: NCT05399251
Title: Relationship Between Serum 1,25-dihydroxy Vitamin D and Markers of Bone Metabolism in Renal Dysfunction Patients
Status: Completed | Type: Observational
Sponsor: Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Zaib Un Nisa Khan, PRINCIPAL INVESTIGATOR, Aga Khan University Hospital, Pakistan
Other Study IDs: ERC # 2020-3295-14097
Record Dates: First submitted 2022-02-14; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Chronic Kidney Disease-Mineral and Bone Disorder
Keywords: renal dysfunction; bone metabolism marker; 1,25(OH)2 vitamin D
MeSH Terms: conditions — Chronic Kidney Disease-Mineral and Bone Disorder; Renal Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This cross-sectional study was conducted, including those subjects tested for 1,25(OH)2D during Jan 2015-Dec 2021. Estimated glomerular filtration rate (eGFR) was calculated and subjects were classified into chronic kidney disease (CKD) stages. Associations between biochemical marker, calcium, phosphorus, magnesium, alkaline phosphatase, 1,25(OH)2D and CKD stages was determined.

ELIGIBILITY:
Inclusion Criteria:

• Data of serum 1,25(OH)2D available

Exclusion Criteria:

• Serum1,25(OH)2D is not available

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Laboratory data of patients tested for 1,25(OH)2D from January 2015 to December 2021 was retrieved from laboratory integrated systems (ILMS), and only the initial results for 1,25(OH)2D were included.
Sampling Method: Non-Probability Sample
Enrollment: 1553 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
concentration of serum 1,25 dihydroxy vitamin D in U/L in five stages of chronic kidney disease | 7 year
  In CKD, 1-alfa-hydroxylase activity in the kidneys is reduced, leading to decreases in the level of the activated form of vitamin D (1,25- dihydroxy vitamin D), resulting in secondary hyperparathyroidism and bone disease. This study aimed to determine the concentration of 1,25 dihydroxy vitamin D in different stages of CKD.
concentration of serum calcium in mg/dl in five stages of chronic kidney disease | 7 years
  in renal tubules, 1,25- dihydroxy vitamin D increase reabsorption of calcium from renal filtrate and thus stabilize blood calcium levels. in CKD, with deterioration of kidney function, stage V, the levels of calcium drops resulting in hypocalcemia.

IPD SHARING:
Plan to Share IPD: No